CLINICAL TRIAL: NCT06344676
Title: Estudi de l'Impacte de la Soledat no Volguda Incorporant un Robot Social en Centres Residencials
Brief Title: Study of the Impact of a Social Robot on Unwanted Loneliness in Elderly People Living in Nursing Homes
Acronym: WITHPEPPER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Domenech (Other)
Responsible Party: Sponsor-Investigator, Sara Domenech, Researcher, Fundacio Salut i Envelliment UAB
Organization: Fundacio Salut i Envelliment UAB (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FSIE2024Robot; 6773 (Other: CERec UAB)
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Elderly People; Nursing Home Residents; Loneliness; Quality of Life; Wellbeing; Social Interaction
Keywords: social robots; loneliness; nursing homes; quality of life; wellbeing
MeSH Terms: interventions — Range of Motion, Articular; Relational Autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): This group will do the usual therapies and activities that were doing before the enrolment in the study
  Interventions: Other: Usual Care
- Robot (Experimental): This group will do the usual therapies and activities that were doing before the enrolment in the study plus:
  * 3 weekly individual cognitive stimulation sessions of 10 minutes.
  * 2 weekly group mobility sessions of 30 minutes.
  * 1 monthly group social session of 60 minutes
  Interventions: Other: Cognitive; Other: Mobility; Other: Social; Other: Relational; Other: Usual Care

INTERVENTIONS:
Other: Cognitive — Tree 10 minutes individual sessions per week involving memory, attention and executive functions tasks.
  Arms: Robot
Other: Mobility — Two 30 minutes group session per week involving physical activity assisted by a social robot.
  Arms: Robot
Other: Social — One 60 minutes group session per month assisted by a social robot that facilitates talking about costumes and traditions.
  Arms: Robot
Other: Relational — Unrestricted individual interaction of the user with the Pepper robot to obtain information of interest for the user (menu, time, date, place and calendar of activities of the residential. center) and 1 individual monthly videoconference with the family of 10 minutes of duration.
  Arms: Robot
Other: Usual Care — Attentions and treatments received by the persons before the enrollment in the study.

SUMMARY:
The goal of this clinical trial is to assess the usefulness of social robots reducing unwanted loneliness in persons over 65 living in nursing homes. The main questions it aims to answer are:

* Can social robots reduce unwanted loneliness?
* Can social robots improve quality of live and well-being? The selected centers are organized in several classes of living units. Living units are independent physical spaces with their own common facilities for the persons living in (usually around 15). Living units of the same class gather persons with similar characteristics.

To compare the added value of the robots half of the living units will be allocated to a control group, and the other half to the intervention group.

The persons in living units allocated to the control group will receive the same attentions and care which were receiving before the enrollment in the study, whereas the persons allocated to the intervention group will add a social robot to their usual therapies and activities. Namely participants will do three weekly individual cognitive stimulation sessions of 10 minutes each one, two weekly group mobility sessions of 30 minutes, one monthly conversational group about customs and traditions of 60 minutes, one 10 minutes videoconference per month with their relatives. Furthermore, participants will be able to interact freely with the robot to obtain information about the center (for instance, what is for dinner) and its activities.

The intervention will last 8 weeks. To assess the effectivity, the investigators will assess both groups, before the intervention, at the end of the intervention and 4 weeks after finishing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* To be 65 years old or older.
* To live indefinitely for more than 6 months in the participating nursing home (to avoid the effect of the adaptation period).
* Provide the informed consent.

Exclusion Criteria:

* Impossibility to understand and/or answer the loneliness questionnaire for themselves.
* To have physical, cognitive or other conditions preventing the use of the robot platform.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Loneliness | weeks 0, 8 and 12
  Change in the UCLA Loneliness Scale (Version 3). The UCLA Loneliness Scale is a 20-item scale (Russell, 1996) that includes statements (e.g., How often do you feel alone?) rated on a four-point Likert scale ranging from 1 (never) to 4 (always). The total score ranges from 20 to 80. Higher scores indicate greater degrees of loneliness.

SECONDARY OUTCOMES:
Well-being | weeks 0, 8 and 12
  Change in the World Health Organisation- Five Well-Being Index (WHO-5).The WHO-5 is a short, self-administered measure of well-being over the last two weeks. It consists of five positively worded items that are rated on 6-point Likert scale, ranging from 0 (at no the time) to 5 (all of the time). The total score ranges from 0 to 100, with lower scores indicating worse well-being.
Quality of life, irrespective of the disease | weeks 0, 8 and 12
  Change in the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L). The EQ-5D-5L can assess patients' quality of life, irrespective of the disease. It covers 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems).
  The descriptive system defines 3,125 distinct health-states. Responses can be combined in a form of a 5-digit number (the best state "11111" meaning no problems at any of dimension to the worst state "55555" meaning unable/extreme problems at all five dimensions). The second part of the instrument is a 20 cm visual analog scale (EQ VAS) ranging from 0 (worst health you can imagine) to 100 (best health you can imagine)
Satisfaction with life | weeks 0, 8 and 12
  Change in the Satisfaction With Life Scale (SWLS). A 5-item scale designed to measure global cognitive judgments of one's life satisfaction (not a measure of either positive or negative affect).
  Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. The five responses are summed to produce a total score for the scale. Total scores can, thus, range from a minimum of 5 to a maximum of 35. Higher scores indicate greater degrees of satisfaction with life.
Depressive symptoms | weeks 0, 8 and 12
  Change in 5-item version of Yesavage's Geriatric Depression Scale (GDS-5). This is useful for identify depressive symptoms among elder people. The presence of 2 or more depressive symptoms is indicative of depression. Higher scores indicate greater degrees of depressive symptoms.
Social Support | weeks 0, 8 and 12
  Change in the Lubben Social Network Scale (LSNS-6). It is a self-report measure of social engagement including family and friends. The total score is calculated by finding the sum of all items. the score ranges between 0 and 30, with a higher score indicating more social engagement
  It is a self-report measure of social engagement including family and friends. The total score is calculated by finding the sum of all items. the score ranges between 0 and 30, with a higher score indicating more social engagement
Communication | weeks 0, 8 and 12
  Change in the Holden Communication Scale (HCS). This is a scale of 12 items rated from 0 to 4 points completed by a professional based on observation of the person with dementia for a certain period of time. It quantifies, based on the degree of deterioration, those aspects that relate the interrelation of the patient with his immediate environment, and the variables refer to observation, knowledge of reality and communication. A higher score indicates greater impairment.

IPD SHARING:
Plan to Share IPD: No
Informed consent states that data will not be used by other persons.